CLINICAL TRIAL: NCT00264290
Title: Valganciclovir to Reduce T Cell Activation in HIV Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H10775-26933-01; SFGH GCRC #976; 5 P30 AI 27763 - Hunt; Roche VAL 104; 5P30AI027763 (NIH)
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Results first posted 2013-11-08 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections; Cytomegalovirus Infections
Keywords: HIV; CMV; T Cell activation; Valganciclovir
MeSH Terms: conditions — HIV Infections; Cytomegalovirus Infections | interventions — Valganciclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Valganciclovir (Experimental): 900mg PO qd
  Interventions: Drug: Valganciclovir
- Placebo (Placebo Comparator): 900mg PO qd
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valganciclovir — 900mg PO qd x 8 weeks followed by 4 weeks of observation on background antiretroviral (ARV) regimen alone.
  Other Names: Valganciclovir (Valcyte); Placebo
  Arms: Valganciclovir
Drug: Placebo — Placebo designed to resemble Valganciclovir
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether treatment with valganciclovir decreases T cell activation levels among HIV-infected patients with asymptomatic cytomegalovirus (CMV) co-infection, potentially improving immune responses to antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Infection with HIV >1 year in duration.
* Age >18
* Cytomegalovirus (CMV) antibody positive.
* All Cluster of Differentiation 4 (CD4)+ T cell counts in the last year and at screening <350 cells/mm3
* On a stable highly addictive antiretroviral therapy (HAART) regimen (DHHS definition) for the preceding 6 months.

  * 90% adherence to antiretroviral therapy within the preceding 30 days.
* Females of childbearing potential must have a negative serum pregnancy test at screening and all subjects must agree to use a double-barrier method of contraception throughout the study period.
* Screening %Cluster of differentiation 38 (CD38)+ Human leukocyte antigen-D-related (HLA-DR)+ Cluster of differentiation 8 (CD8)+ T cells >10%

Exclusion Criteria:

* Patients intending to modify antiretroviral therapy in the next 16 weeks.
* Serious illness requiring hospitalization or parental antibiotics within preceding 3 months.
* Evidence of active symptomatic CMV end-organ disease.
* Treatment with valganciclovir or ganciclovir in the past 30 days.
* Concurrent treatment with immunomodulatory drugs.
* Concurrent treatment with nephrotoxic drugs
* Screening absolute neutrophil count <1,000 cells/mm3, platelet count <100,000 cells/mm3, hemoglobin < 8mg/dL, estimated creatinine clearance <50 mL/minute.
* Men who are considering having children will also be excluded given potential effects of valganciclovir on spermatogenesis.
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-08; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter W. Hunt, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital - General Clinical Research Center, San Francisco, California, United States

REFERENCES:
- [Background] Hunt PW, Martin JN, Sinclair E, Bredt B, Hagos E, Lampiris H, Deeks SG. T cell activation is associated with lower CD4+ T cell gains in human immunodeficiency virus-infected patients with sustained viral suppression during antiretroviral therapy. J Infect Dis. 2003 May 15;187(10):1534-43. doi: 10.1086/374786. Epub 2003 Apr 23. PMID 12721933
- [Result] Hunt PW, Martin JN, Sinclair E, Epling L, Teague J, Jacobson MA, Tracy RP, Corey L, Deeks SG. Valganciclovir reduces T cell activation in HIV-infected individuals with incomplete CD4+ T cell recovery on antiretroviral therapy. J Infect Dis. 2011 May 15;203(10):1474-83. doi: 10.1093/infdis/jir060. PMID 21502083

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cytomegalovirus (CMV)-seropositive adults with chronic HIV infection were recruited at one US clinical site.
Pre-assignment Details: Of 60 screened subjects, 3 refused participation and 27 did not meet eligibility criteria. The most common reason for exclusion was <10% activated Cluster of differentiation * (CD8)+ T cells.
Groups:
- Placebo: Placebo PO qd x 8 weeks followed by 4 weeks of observation on background antiretroviral (ARV) regimen alone.
- Valganciclovir: 900mg PO qd
  Valganciclovir : 900mg PO qd x 8 weeks followed by 4 weeks of observation on background antiretroviral (ARV) regimen alone.
Period: Intervention (8 Weeks)
Arm/Group | Placebo | Valganciclovir
Started | 16 | 14
Completed | 15 | 14
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Observation (4 Weeks)
Arm/Group | Placebo | Valganciclovir
Started | 15 | 14
Completed | 15 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo PO qd x 8 weeks followed by 4 weeks of observation on background ARV regimen alone.
- Valganciclovir: 900mg PO qd
  Valganciclovir : 900mg PO qd x 8 weeks followed by 4 weeks of observation on background ARV regimen alone.
- Total: Total of all reporting groups
Arm/Group | Placebo | Valganciclovir | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 50 [44 to 59] | 48 [43 to 55] | 49 [43 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 16 | 12 | 28
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in %CD38+ Human Leukocyte Antigen-D-related (HLA-DR)+ CD8+ T Cells From Baseline to Week 8.
Description: The percentage of activated (CD38+ HLA-DR+) CD8+ T cells was measured on fresh whole blood at screening/baseline. T cell activation was measured on peripheral blood mononuclear cells (PBMCs)in batch at the end of the study.
Time Frame: Baseline, 8 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of activated T cells
Arm/Group | Placebo | Valganciclovir
Number analyzed (Participants) | 15 | 14
percentage of activated T cells | 1.3 [-2.6 to 5.8] | -4.0 [-5.7 to -0.9]

2. Secondary Outcome: Change in CMV DNA Shedding From Baseline to Week 8.
Description: Change in percentage of participants with detectable CMV DNA. Herpesvirus DNA levels were assessed by polymerase chain reaction (lower limit of detection, 150 copies/mL) on saliva and seminal plasma.
Time Frame: baseline and week 8
Measure: Number; unit: percentage of participants
Arm/Group | Valganciclovir | Placebo
Number analyzed (Participants) | 14 | 16
percentage of participants | -36 | 0
Statistical Analysis 1: Comparison: Valganciclovir vs Placebo; Test type: Other; p = 0.007, Fisher Exact

3. Secondary Outcome: Change in Cluster of Differentiation 4 (CD4) Counts at Week 8
Time Frame: Baseline and week 8
Measure: Mean (95% Confidence Interval); unit: CD4 cells/mm3
Arm/Group | Placebo | Valganciclovir
Number analyzed (Participants) | 16 | 14
CD4 cells/mm3 | -1 [-19 to 16] | -8 [-38 to 22]

4. Secondary Outcome: Change in Percent of CD38+HLA-DR+ CD8+ T Cells After a 4-week Washout Period
Description: Change from baseline at week 12
Time Frame: Baseline and Week 12
Measure: Mean (95% Confidence Interval); unit: %CD38+HLA-DR+ CD8+ T cells
Arm/Group | Placebo | Valganciclovir
Number analyzed (Participants) | 16 | 14
%CD38+HLA-DR+ CD8+ T cells | 1 [-3 to 5] | -4.1 [-6.8 to -1.1]

5. Secondary Outcome: Number of Participants With Positive CMV DNA After a 4-week Washout Period
Description: Number of Participants with positive CMV DNA at any site at week 12
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Valganciclovir
Number analyzed (Participants) | 16 | 14
Participants | 0 | 3

6. Secondary Outcome: Change in CD4 Counts After a 4-week Washout Period
Description: Change from baseline at week 12
Time Frame: Week 12
Measure: Mean (95% Confidence Interval); unit: cells/mm3
Arm/Group | Placebo | Valganciclovir
Number analyzed (Participants) | 16 | 14
cells/mm3 | 6 [-11 to 23] | -17 [-47 to 12]

ADVERSE EVENTS:
Time Frame: 8 weeks of study treatment and a 4-week Observation Period
Arm/Group | Placebo | Valganciclovir
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | Valganciclovir (N=14)
congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes